CLINICAL TRIAL: NCT02995707
Title: The Phase II Clinical Trials of Thalidomide in NTDT
Brief Title: The Effective and Safety of Thalidomide in NTDT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiao-Lin Yin (Other)
Responsible Party: Sponsor-Investigator, Xiao-Lin Yin, Director, NO.3 Hospital of the People's Liberation Army, 303rd Hospital of the People's Liberation Army
Organization: 303rd Hospital of the People's Liberation Army (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303PLA
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Thalassemia
Keywords: Thalidomide NTDT
MeSH Terms: conditions — Thalassemia | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thalidomide thalassemia (Experimental): thalidomide:50mg/d p.o
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — thalidomide:50mg/d p.o at bedtime
  Other Names: fǎn yìng tíng

SUMMARY:
This is an exploratory experiment, aims to explore the effective and safety of thalidomide in the treatment of NTDT to improve the hemoglobin level, improve the quality of life, reduce blood transfusion, so as to avoid the adverse reactions caused by transfusion.15~30 patients will be enrolled, including type α 5~13 cases, type β 10~17 cases.

DETAILED DESCRIPTION:
The project is a single arm research of thalidomide in NTDT,patients volunteered to participate in this trial and met the following inclusion criteria will be enrolled: age from 18~65, Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less. Subjects should take thalidomide 50mg per day for 12 weeks. During this time, hepatic and renal function, hematologic function, electrocardiogram and the adverse reactions were closely observed. According to the protocol, the blood routine, peripheral blood reticulocyte count, nucleated red blood cell count, hemoglobin electrophoresis and other indicators were evaluated in screening-period visit, 4-weeks visit, 8-weeks visit and 12-weeks visit.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be considered for admission to the trial:

* Diagnosis of NTDT;
* Ages 18-65 years;
* ECOG: 0~2 scores;
* Sign an informed consent agreeing to the clinical trial participation.

Exclusion Criteria:

Patients presenting with any of the following criteria will not be included in the trial:

* Patients received hydroxycarbamide, Yisui Shengxue Granule in three months;
* Women during Pregnancy, breastfeeding or those of childbearing age who do not want to take contraceptive measures;
* Patients had comorbidities like severe heart or lung diseases, liver dysfunction, cerebrovascular, cardiovascular, liver, kidney, tumor or other serious primary diseases;
* Patients Allergic to the drug ingredients;
* Patients with any Mental problem;
* Patients had Participated in other drug clinical trials in the past 1 month;
* Patients had a history of venous or arterial thrombosis;
* In certain circumstances that the researchers determined it was not suitable for the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The level of Hemoglobin | 18 months
  All participants will complete the treatment for 18 months, the hemoglobin levels will be observed during the treatment.

SECONDARY OUTCOMES:
The effects of relative and absolute values of HbF | 18 months
  The highest hemoglobin value will be observed,the value increased more than 20g/L defined as the marked effect, increased to 10~20g/L defined as effective, otherwise invalid.

CONTACTS AND LOCATIONS:
Overall Officials: Yin X Lin, director, Study Director — NO.3 Hospital of the Chinese People's Liberation Army
Locations (1):
- NO.3 Hospital of the Chinese People's Liberation Army, Nanjing, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Three months later after the last visit，summery report will be shared with other researchers through database.

REFERENCES:
- [Derived] Ren Q, Zhou YL, Wang L, Chen YS, Ma YN, Li PP, Yin XL. Clinical trial on the effects of thalidomide on hemoglobin synthesis in patients with moderate thalassemia intermedia. Ann Hematol. 2018 Oct;97(10):1933-1939. doi: 10.1007/s00277-018-3395-5. Epub 2018 Jun 22. PMID 29931453